CLINICAL TRIAL: NCT00973310
Title: A Phase II Study on the Safety and Efficacy of Radiation Therapy and Concurrent Erlotinib in Locally Advanced Non-small-cell Lung Cancer
Brief Title: Erlotinib Concurrent With Radiation Therapy in Non-small-cell Lung Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TMU-CIH-L001
Record Dates: First submitted 2009-09-08; First posted 2009-09-09 (Estimated); Last update posted 2015-12-22 (Estimated); Status verified 2010-12

CONDITIONS: Carcinoma, Non-Small Cell Lung
Keywords: Non-small-cell lung cancer; Radiation therapy; Epidermal growth factor receptor; Tyrosine kinase inhibitor
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Radiotherapy; Erlotinib Hydrochloride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Combined Treatment arm (Experimental): All the patients received oral erlotinib and concurrent radiation therapy
  Interventions: Other: Radiation Therapy and EGFR-TKI target therapy

INTERVENTIONS:
Other: Radiation Therapy and EGFR-TKI target therapy — Patients with locally advanced NSCLC received oral erlotinib (150 mg, qd) for about 6-7 weeks during the course of radiation therapy (60-70Gy in a fraction dose of 2 Gy, 5 fractions per week)
  Other Names: Tarceva, Radiotherapy

SUMMARY:
The purpose of this study is to determine the safety and efficacy of the concurrent use of erlotinib and radiation therapy in the treatment of locally advanced non-small lung cancer.

DETAILED DESCRIPTION:
Non-small cell lung cancer (NSCLC) is still the leading cause of cancer death world-wide. Radiation therapy (RT) is one of the most important treatment choices in locally advanced NSCLC. Combination of RT and chemotherapy could improve treatment outcomes. However, the combined modality could not be used in many patients due to severe toxicities. EGFR-TKI shows great efficacy in the treatment of NSCLC, and many phase I/II studies established its safety in combination with RT. This phase II study is to further evaluate the efficacy and safety of the combination of RT and erlotinib in the treatment of locally advanced NSCLC. Eligible patients include patients with stage IIIA/IIIB NSCLC, who are not suitable for or refused to receive concurrent chemoradiotherapy. Eligible patients will receive oral erlotinib (150mg qd)throughout the course of thoracic RT (60-70 Gy). The primary endpoint is progression free survival and the second endpoints are overall survival and any grade III and above toxicities. We are going to recruit 50 patients for this study.

ELIGIBILITY:
Inclusion Criteria:

* Aged 18-70 years，
* Patients with stage IIIA-IIIB NSCLC
* adequate hematologic (WBC and platelet counts within normal limits), hepatic (total bilirubin level <= two times the upper limit of normal), and renal (creatinine clearance >= 50mL/min) functions
* No history of chemotherapy or less than 4 cycles neoadjuvant chemotherapy
* Can not tolerate or refuse concurrent chemoradiotherapy
* No history of thoracic RT
* Written informed consent obtained

Exclusion Criteria:

* With other malignancy
* With severe cardiopulmonary disease
* Compromised liver or renal function that could not tolerate the combined therapy
* Received thoracic RT before
* Pregnant or breast-feeding women
* Present with active infection
* Uncontrolled diabetes
* Concurrent use of other anti-cancer agents

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2009-10; Primary Completion 2016-11 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Evidence of clinically definite disease progression | 3 year

SECONDARY OUTCOMES:
All cause mortality and any grade III and above toxicities | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Zhiyong Yuan, M.D., Ph.D., Principal Investigator — Tianjin Medical University Cancer Institute and Hospital
Locations (1):
- Tianjin Medical University Cancer Institute and Hospital, Tianjin Key Laboratory of Cancer Prevention and Therapy, Tianjin, Tianjin Municipality, China

REFERENCES:
- [Derived] Zhuang H, Hou H, Yuan Z, Wang J, Pang Q, Zhao L, Wang P. Preliminary analysis of the risk factors for radiation pneumonitis in patients with non-small-cell lung cancer treated with concurrent erlotinib and thoracic radiotherapy. Onco Targets Ther. 2014 May 24;7:807-13. doi: 10.2147/OTT.S62707. eCollection 2014. PMID 24920921